CLINICAL TRIAL: NCT06341699
Title: Studio Del Milieu Steroideo in Pazienti Obesi
Brief Title: Study of the Steroid Hormone Milieu in Obese Patients
Acronym: MiSterO
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: 05C308
Record Dates: First submitted 2024-03-16; First posted 2024-04-02 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Obesity, Morbid
Keywords: hypercortisolism; hypogonadism
MeSH Terms: conditions — Obesity, Morbid; Cushing Syndrome; Hypogonadism

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples for DNA analysis to study polymorphisms of glucocorticoid and androgen receptors, and NGS to look for rare variants in genes associated with hypogonadotropic hypogonadism and hypercortisolism.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to evaluate the actual secretion of cortisol and testosterone in obese male subjects, together with the receptor sensitivity to these hormones in order to understand whether the hormonal milieu deriving from these parameters is associated with alterations in bone metabolism, lipoprotein concentration and function, and/or the severity and complications of obesity.

It will be also investigated if this hormonal milieu is a predictive factor for cardiovascular disease in obese patients.

Eligible subjects are male patients (age 18-80 years) with severe obesity and no other known causes of hypercortisolism or hypogonadism.

Questionnaires for the evaluation of mood and symptoms will be collected upon enrollment, patient's anamnestic and clinical data relating to disease complications, BMI, previous blood tests, cortisol suppression with dexamethasone 1 mg will be collected, and blood sample will be sent to and analyzed at a centralized laboratory for the study of Steroid hormones, bone metabolism, lipoprotein function, genetics and receptor analysis.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity

Exclusion Criteria:

* patients suffering from severe systemic pathologies, fever, chronic inflammatory states known to cause PCR >10 mg/dL
* use of corticosteroids at the time of enrollment
* the patient's poor understanding of spoken and written Italian
* patients suffering from primary pathologies of the testicle, known at enrollment
* patients suffering from hypothalamic-pituitary or adrenal pathologies already known at the time of enrollment

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected with severe obesity
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Association of androgen milieu with the severity of obesity | 2024
  Evaluate the association of hypogonadism and/or androgen receptor polymorphisms that reduce sensitivity to androgens with: patients' BMI; comorbidities of obesity, and bone metabolism
Association of cortisol milieu with the severity of obesity | 2024
  Evaluate the association of hypercortisolism and/or glucocorticoid receptor polymorphisms that increase sensitivity to cortisol with: patients' BMI; comorbidities of obesity, and bone metabolism
Algorithm fo CV risk in obesity | 2024
  Use of artificial intelligence methods to hypothesize an algorithm including steroid milieu that can identify obese patients at greater cardiovascular risk

SECONDARY OUTCOMES:
Prevalence of hypogonadism in morbid obesity | 2024
  To evaluate the prevalence of hypogonadism in patients with severe obesity using EMAS criteria
Prevalence of patients with morbid obesity unresponsive to overnight suppression test | 2024
  To evaluate the prevalence of patients with severe obesity positive to Nugent testing
Enrichment in rare HH variants in obese patients with central hypogonadism | 2025
  Compare the enrichment in rare variants for HH-associated genes in obese patients with hypogonadotropic hypogonadism, compared to the general population
Enrichment in rare variants associated with hypercortisolism in obese patients unresponsive to Nugent testing | 2025
  Compare the enrichment in rare variants in genes associated with hypercortisolism in obese patients unresponsive to Nugent testing, compared to the general population

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxlogico Italiano, Hospital San Giuseppe, Piancavallo, Oggebbio, Verbania, Italy